CLINICAL TRIAL: NCT05998746
Title: Comparison of ASA and CFS in Predicting Peri- and Postoperative Outcomes in Elective Patients Older Than 65 Years
Brief Title: Comparison of ASA and CFS in Anesthesiology
Acronym: CACA
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: Osijek University Hospital (Other)
Responsible Party: Sponsor
Other Study IDs: OS-UH23
Record Dates: First submitted 2023-08-11; First posted 2023-08-21 (Actual); Last update posted 2023-08-21 (Actual); Status verified 2023-08

CONDITIONS: Frailty
Keywords: American Society of Anesthesiologists physical status;; Clinical frailty; Elderly; Treatment outcome
MeSH Terms: conditions — Frailty

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Patient Registry: Yes
Target Follow-Up Duration: 2 Months
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

SUMMARY:
In addition to the regular ASA classification, patients would also be assigned the Clinical frailty scale (CFS) during preoperative examinations in anesthesiology clinics. The aim is to compare the usefulness of ASA and CFS categorization for predicting perioperative and postoperative complications and length of postoperative stay in elective surgeries.

DETAILED DESCRIPTION:
CFS significantly correlates with complications in patients treated in emergency department. This study is expected to provide information on how CFS correlates with complications and length of stay in elective surgeries.

In addition to the regular ASA classification, patients would also be assigned the Clinical frailty scale (CFS) during preoperative examinations in anesthesiology clinics.

The respondents are all elective patients over 65 years of age who have not had previously recorded mental difficulties that interfere with their daily life. Patients suffering from senile dementia would not be excluded from this study.

After the treatment was completed, the medical history of each patient would be reviewed and statistically processed.

The aim is to compare the usefulness of ASA and CFS categorization for predicting perioperative and postoperative complications and length of postoperative stay in elective surgeries.

ELIGIBILITY:
Inclusion Criteria:

* All elective patients older then 65 years

Exclusion Criteria:

* Earlier mental difficulties that affect everyday life, senile dementia is not exclusion criteria

Min Age: 65 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Older Adult
Study Population: Study population is all elective patients of the Osijek University Hospital older then 65 years who were included during the preoperative examination.
Sampling Method: Non-Probability Sample
Enrollment: 200 (Estimated)
Dates: Start 2023-07-17 (Actual); Primary Completion 2024-04-30 (Estimated); Study Completion 2024-06-03 (Estimated)

PRIMARY OUTCOMES:
Peri- and postoperative complications | During 2 months after elective operation
  Peri- and postoperative complications depending on CFS and ASA

SECONDARY OUTCOMES:
Length of stay in hospital | During 2 months after elective operation
  Length of stay in hospital after elective operation depending on CFS and ASA

CONTACTS AND LOCATIONS:
Overall Officials: Slavica Kvolik, MD, Study Chair — Osijek University Hospital; Medical Faculty Osijek
Locations (1):
- University Hospital Centre Osijek, Osijek, Croatia